CLINICAL TRIAL: NCT02623764
Title: EEG-cholinergic Index and Its Validation of Clinical Response to Treatment With Cholinesterase Inhibitors
Brief Title: EEG-cholinergic Index and Clinical Response to Treatment With Cholinesterase Inhibitors
Acronym: Cholindex
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Landspitali University Hospital (Other)
Collaborators: Mentis Cura (Industry)
Responsible Party: Sponsor
Other Study IDs: LSH-15-002
Record Dates: First submitted 2015-11-05; First posted 2015-12-08 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer´s Disease
Keywords: Alzheimer´s disease; Lewy body dementia; Parkinson dementia; EEG; Cholinergic index
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- MCI due to Alzheimer´s disease: Individuals with MCI diagnosed with Alzheimer´s disease on the basis of cognitive decline and positive biomarkers by MRI and/or Cerebro Spinal Fluid (CSF) analysis. The intervention is donepezil in recommended doses, 5mg/day for a month and then 10mg/day. Cholinergic index in EEG will be measured before initiating treatment, after 3 and 6 months and related to clinical response of treatment
- Mild dementia due to Alzheimer´s disease: Individuals with mild dementia and diagnosed with Alzheimer´s disease on the basis of cognitive decline and positive biomarkers by MRI and/or CSF analysis. The intervention is donepezil in recommended doses, 5mg/day for a month and then 10mg/day. Cholinergic index in EEG will be measured before initiating treatment, after 3 and 6 months and related to clinical response of treatment
- Mild dementia due to Lewy body disease: Individuals with mild Lewy body dementia. The intervention is Exelon patches in recommended doses, 4.6mg/day for a month and then 9.5mg/day. Cholinergic index in EEG will be measured before initiating treatment, after 3 and 6 months and related to clinical response of treatment

SUMMARY:
Drug treatment with cholinesterase inhibitors is indicated for treatment of Alzheimer´s disease and in most cases, one of these drugs is prescribed as soon as the diagnosis has been made. Nevertheless, it has been shown in several studies that up to 30% of patients do not benefit from treatment. These drugs can have side effects, most frequently from the gastrointestinal tract with nausea, diarrhea and discomfort in the abdomen as the most frequent signs. It is therefore important to know before the treatment is initiated if the patient will likely benefit from the drug or not. It is not possible today with current knowledge but this project aims to evaluate a specific index, calculated from an EEG registration (the EEG-cholinergic index) for this purpose. A conventional EEG registration is done before treatment and the cholinergic index calculated from the EEG registration is compared to the clinical outcome. The duration of follow up is 6 months with an extension of further 6 months.

DETAILED DESCRIPTION:
Patients will be recruited in a Memory Clinic. Three possible groups of participants will be offered participation:

* Those with Mild Cognitive Impairment (MCI) but with biomarkers of Alzheimer´s disease (AD) that are conclusive enough to lead to the diagnosis of AD and to initiate medical treatment.
* Those with early dementia of AD that are offered medical treatment and are able to give consent.
* Those with early dementia of Lewy body dementia or Parkinson dementia that are offered medical treatment.

All eligible participants are evaluated by the Mini Mental State Examination (MMSE), Consortium to Establish Registry in Alzheimer´s Disease (CERAD 10 word test; working memory, delayed memory and recognition) and Clock Drawing Test (CDT). In addition, the Addenbrooke test will be used.

Patients with AD irrespective of stage will be offered treatment with donepezil, the most used and cheapest cholinesterase inhibitor in Iceland. The dosis will be as usual, 5mg in the evening for four weeks, then increased to 10mg in the evening.

Patients with Lewy body dementia and Parkinson dementia are offered rivastigmine in patch as this is the only medication with the indication of cognitive impairment in these disorders. The starting dose is 4.6mg/day increased to 9.5mg/day after 4 weeks.

After 3 months, each participant is evaluated again with the same tests as before initiating treatment (continuous variables). The clinical effect is also rated according to Clinical Dementia Rating (CDR; categorical variables). An EEG registration is performed. Adherence to drug therapy as well as evaluation of side effects is registrated.

After 6 months, each participant is evaluated again as after 3 months. This is the primary end point.

After 12 months an additional evaluation is performed by the same instruments (secondary endpoint).

The EEG is thus registrated 3 times (primary end point) or 4 times (secondary end point as the first registration was done during the diagnostic work up before entering the project. The EEG will reveal group wise category (Normal, AD or Lewy according to the third edition (SIGLA) of Mentis Cura). An analysis of the cholinergic index is not revealed to the clinician that is thus blinded to this part of the EEG analysis.

The project will be analysed based on all available information after primary end point. A second analysis will be performed after the second end point.

ELIGIBILITY:
Inclusion Criteria:

* Mild Cognitive Impairment or mild dementia due to Alzheimer´s disease or with dementia due to Lewy body disease.

Exclusion Criteria:

* Too advanced dementia (5 or more on Global Deterioration Scale)
* likelihood of poor compliance due to social circumstances, drug or alcohol abuse or other defined causes.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed at a Memory Clinic with Mild Cognitive Impairment or mild dementia due to Alzheimer´s disease or with dementia due to Lewy body disease
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2015-12; Primary Completion 2019-05 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Addenbrooke cognitive battery at 3 months and at 6 months | Baseline, 3 months, 6 months
  Addenbrooke cognitive battery will be used before initiating treatment (baseline), after 3 months and after 6 months

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE) | Baseline, 3 months, 6 months
  MMSE will be used before initiating treatment (baseline), after 3 months and after 6 months
CERAD-10 word test | Baseline, 3 months, 6 months
  CERAD-10 word test will be used before initiating treatment (baseline) after 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jon Snaedal, MD, Principal Investigator — Professor